CLINICAL TRIAL: NCT02740218
Title: APPRECIATE (Apremilast Clinical Treatment Experience in Psoriasis): A Multi-center, Retrospective Observational Study of Real-World Experience of Psoriasis Patients Treated With Apremilast in Clinical Dermatology Practice
Brief Title: A Study of Real-World Experience of Psoriasis Patients Treated With Apremilast in Clinical Dermatology Practice
Acronym: APPRECIATE
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSOR-013
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; Apremilast; APPRECIATE; Dermatology; Retrospective; Observational
MeSH Terms: conditions — Psoriasis | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Psoriasis patients: Single cohort of psoriasis patients treated with OTEZLA (apremilast)
  Interventions: Other: Patient questionnaire

INTERVENTIONS:
Other: Patient questionnaire — Patients will be asked to complete a questionnaire regarding their expectations, experience and satisfaction in taking OTEZLA (apremilast) treatment

SUMMARY:
This is a retrospective, multi-center observational cohort study. This study will be implemented first in Germany (approximately 50 sites), the United Kingdom (approximately 20 sites) and Sweden (approximately 25 sites), followed by a selected number of countries in Europe, depending on apremilast local availability. The design of this apremilast retrospective study aims to provide clinical information regarding the treatment initiation and outcomes in psoriasis patients when prescribed apremilast in real world settings. In addition, this study is aiming at capturing physicians' and patients' treatment goals when initiating apremilast and whether these goals are achieved following apremilast use. This study is primarily descriptive in nature, and no a priori hypotheses are specified. Patients must voluntarily sign an informed consent form, be 18 or over, have been diagnosed with plaque psoriasis and have been treated with apremilast during the previous 5-7 months to participate in this study. They must not be involved in any other clinical study involving apremilast.

ELIGIBILITY:
Inclusion Criteria:

1. Must have understood and voluntarily signed the Informed Consent Form (ICF).
2. Age ≥ 18 years at the time of signing the ICF.
3. Diagnosed with plaque psoriasis.
4. Initiated treatment with apremilast 6 months (+/- 1 month) previously (patients may or may not have completed 6 months of apremilast treatment)

Exclusion Criteria:

1. Refusal to participate in this study or current participation in the treatment phase of an interventional clinical trial.
2. Started apremilast as part of a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient charts will be selected for data abstraction by participating dermatologists and will be determined eligible for study enrollment based on the inclusion criteria. All consecutive adult psoriasis patients who can be contacted 6 months (+/- 1 month) following initiation of treatment with apremilast will be approached for entry to minimize bias in patient selection. All eligible patients will be included in consecutive order regarding the date of the signed Informed Consent.
Sampling Method: Non-Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
The Patient Benefit Index (PBI) outcome score | Up to approximately 7 months
  Is a questionnaire regarding patient expectations and benefit of psoriasis treatment with apremilast, eg, effect on specific symptoms.

SECONDARY OUTCOMES:
Treatment Satisfaction Questionnaire for Medication (TSQM) outcome score | Up to approximately 7 months
  The TSQM-9 is a self-administrated instrument to understand a subject's satisfaction on the current therapy
Percentage of patients achieving PASI75 | Up to approximately 7 months
  PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 16. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The PASI score was set to missing if any severity score or degree of involvement is missing.
Percentages of patients achieving PASI50 | Up to approximately 7 months
  PASI score is based on an assessment of erythema (reddening), induration (plaque thickness), desquamation (scaling), and the percent area affected as observed on the day of examination.
Mean change in Dermatology Life Quality Index (DLQI) | Up to approximately 7 months
  DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the participant is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score is derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
Percentages of patients achieving ≥5 point improvement in DLQI | Up to approximately 7 months
  DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the participant is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score is derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
Percentages of patients achieving PASI50 plus ≥5 point improvement in DLQI | Up to approximately 7 months
  PASI score is based on an assessment of erythema (reddening), induration (plaque thickness), desquamation (scaling), and the percent area affected as observed on the day of examination.
  DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease
Mean change in Body Surface Area (BSA) | Up to approximately 7 months
  BSA was a measurement of involved skin. The overall BSA affected by psoriasis was estimated based on the palm area of the participant's hand (entire palmar surface or "handprint" including the fingers), which equates to approximately 1% of total body surface area.
Mean change in PGA | Up to approximately 7 months
  The PGA is a 5-point scale ranging from 0 (clear) to 4 (severe), incorporating an assessment of the severity of the 3 primary signs of the disease: erythema, scaling and plaque elevation. When making the assessment of overall severity, the assessor factors in areas that have already cleared (ie, have scores of 0) and not just remaining lesions for severity, ie, the severity of each sign was to be averaged across all areas of involvement, including cleared lesions
Percentage of patients achieving PGA 0/1 (clear/almost clear) | Up to approximately 7 months
  The PGA is a 5-point scale ranging from 0 (clear) to 4 (severe), incorporating an assessment of the severity of the 3 primary signs of the disease: erythema, scaling and plaque elevation. When making the assessment of overall severity, the assessor factors in areas that have already cleared (ie, have scores of 0) and not just remaining lesions for severity, ie, the severity of each sign was to be averaged across all areas of involvement, including cleared lesions
Adverse Events (AEs) | Up to approximately 7 months
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (133):
- Austria (17):
  - Medizinische Universität Graz, Graz
  - Praxis Dr. Wolfgang Fuchs, Grosswarasdorf
  - Praxis Dr. Schicher, Klagenfurt
  - Praxis Dr. Wilhelm, Landeck
  - Kepler Universitätsklinikum, Linz
  - Praxis Dr. Dunst-Huemer, Linz
  - Krankenanstalt Rudolfstiftung, Vienna
  - Medizinische Universität Wien, Vienna
  - Praxis Dr. Göttfried, Vienna
  - Praxis Dr. Holub-Hoberger, Vienna
  - Krankenhaus Hietzing, Vienna
  - Praxis Dr. Nordberg, Vienna
  - Praxis Dr. Menzinger, Vienna
  - Praxis Dr. Sator, Vienna
  - Praxis Dr. Perl-Convalexius, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Croatia (5):
  - Klinički bolnički centar Osijek Zavod za dermatologiju i venerologiju, Osijek
  - Klinički bolnički centar Rijeka Klinika za dermatovenerologiju, Rijeka
  - Klinički bolnički centar Split Klinika za kožne i spolne bolesti, Split
  - Klinički bolnički centar Sestre milosrdnice Klinika za kožne i spolne bolest, Zagreb
  - Klinički bolnički centar Zagreb Klinika za dermatovenerologiju, Zagreb
- Czechia (7):
  - Fakultní nemocnice Hradec Králové Klinika nemocí kožních a pohlavních, Hradec Králové, Novy Hradec Králové
  - Nemocnice Pardubického kraje, Pardubice, Pardubice IV
  - Sanatorium profesora Arenberger, Prague, Praha 1
  - Všeobecná fakultní nemocnice v Praze, Prague, Praha 2
  - Fakultní nemocnice v Motole, Prague, Praha 5
  - Nemocnice Jihlava příspěvková organizace, Jihlava
  - FN Plzen Bory Dermatovenerologické oddělení, Pilsen
- Germany (49):
  - Company for Medical Study & Service, Selters, Westerwald
  - Praxis Dr. Harst, Aachen
  - Praxis Dr. Wagner-Schiffler, Aachen
  - Praxis Dr. Dietz, Ampfing
  - Praxis Dr. Bell, Andernach
  - Licca Clinical Research Institute, Augsburg
  - Gefäß- und Hautzentrum Blaustein, Blaustein
  - St. Josef und St. Elisabeth Hospital gGmbH, Bochum
  - Rheinische Friedrich-Wilhelms-Universität Bonn, Bonn
  - Praxis Dr. Jordan, Brühl
  - Elbe Klinikum Buxtehude, Buxtehude
  - Praxis Dr. Schneider, Dachau
  - Praxis Dr. Thelen, Delmenhorst
  - Klinikum Dortmund, Dortmund
  - Praxis Dr. Scheibner, Dresden
  - Praxis Dr. Korge, Düren
  - Praxis für Dermatologie und Venerologie, Allergologie, Eltville
  - Praxis Dr. Schurhammer-Fuhrmann, Endingen
  - Uniklinikum Erlangen, Erlangen
  - Praxis Dr. Huerkamp, Euskirchen
  - Praxis Dr. Swirski, Euskirchen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Praxis Dr. Kämmerer, Freiberg
  - Praxis Dr. Kurzen, Freising
  - GP Dr. Rotterdam & Kollegen, Gelsenkirchen
  - Praxis Dr. med W. Klövekorn, Dr. med. A. Tepe, Dr. med. O. Wilde, Gilching
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Praxis Dr. Schmidt, Kusel
  - Praxis Birgit Zimmermann, Malchow
  - Praxis Dr. Piontek, Mechernich
  - Dermatologische Praxis Dr. med. Schwinn, Memmingen
  - Praxis Büchler, Memmingen
  - Praxis Dr. Antal, Mühldorf
  - Praxis Dr. Cords, Mühlheim
  - Praxis Dr. Liebich, München
  - Technische Universität München, München
  - Universitätsklinikum Regensburg, Regensburg
  - Praxis Dr. Prell, Rosenheim
  - Praxis Dr. Blank, Rostock
  - Praxis Dr. Hoene, Rostock
  - Praxis Dr. Schenkelberger, Sankt Ingbert
  - Praxis Dr. Neisius, Stolberg
  - Praxis Dr. Steinborn, Straubing
  - Universitätsklinikum Tübingen, Tübingen
  - Gemeinschaftspraxis Dr. Christian Fischer, Florian Kreuziger, Vilshofen
  - Praxis Dr. Dehmel, Wasserburg am Inn
  - Praxis Dr. Schmeel, Wesseling
  - Praxis Dr. Buttgereit, Wildau
  - Praxis Dr. Süß, Wittlich
- Ireland (3):
  - Bon Secours Hospital, Tralee, County Kerry
  - Mater Misericordiae University Hospital, Dublin
  - University Hospital Galway, Galway
- Uniiverzitetni klinični center Maribor Oddelek za kožne in spolne bolezni, Maribor, Slovenia
- Spain (4):
  - Hospital Fundacion Alcorcon, Madrid, Alcorcón, Madrid
  - Vithas Xanit Iinternational Hospital, Benalmádena
  - Hospital Universitario San Cecilio (PTS), Granada
  - Hospital Virgen de la Victoria, Málaga
- Sweden (16):
  - Hudkliniken Mälarsjukhuset, Eskilstuna
  - Hudkliniken SU/ Sahlgrenska, Gothenburg
  - Hudmottagningen Karlskoga Lasarett, Karlskoga
  - Hudmottagningen Lindesbergs Lasarett, Lindesberg
  - Capio Citykliniken Lund, Lund
  - Diagnostiskt Centrum Hud Malmö, Malmo
  - SUS Malmö Hudkliniken, Malmo
  - Hudkliniken Vrinnevisjukhuset Norrköping, Norrköping
  - Diagnostiskt Centrum Hud Stockholm, Stockholm
  - Cutisgruppen/Stockholm Hud, Stockholm
  - Hudkliniken SÖS, Stockholm
  - Hudcentrum Hagastaden, Stockholm
  - Karolinska Psoriasis Center, Stockholm
  - Hudkliniken Danderyds Sjukhus, Stockholm
  - Hudmottagningen Trelleborg, Trelleborg
  - Hudmottagningen Västervik, Västervik
- Switzerland (18):
  - Dermatologie Aesche, Basel
  - Somamedica, Basel
  - Ospedale Bellinzona e Valli EOC, Bellinzona
  - Insel Gruppe AG, Bern
  - Clinique dermatologie du Seujet, Geneva
  - Hautarzt Oberaargau AG, Herzogenbuchsee
  - Centre hospitalier universitaire Vaudois (CHUV), Lausanne
  - Studio medico Dr. Pelloni, Lugano
  - Practice Dr. Niklaus, Martigny-Ville
  - Pallas Klinik Olten, Olten
  - Haut und Laserzentrum Dr. Zuder, Sankt Gallen
  - Praxis Dr. med. Christian Schuster, Sankt Gallen
  - Haut und Allergiezentrum Brunnehof, Uster
  - Dr. Tomi Haut- und Laserzentrum, Weinfelden
  - Hautpraxis Dermateam, Winterthur
  - Praxisgemeinschaft Bünz AG, Wohlen
  - Zug Hautarzt, Zug
  - Universitätsspital Zürich, Zurich
- United Kingdom (13):
  - Aberdeen Royal Infirmary, Aberdeen
  - Bradford Teaching Hospitals NHS, Bradford
  - West Suffolk NHS Foundation, Bury St Edmunds
  - East Kent & Canterbury Hospital, Canterbury
  - NHS Dumfries and Galloway, Dumfries
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - West Middlesex University Hospital, Isleworth
  - Chapel Allerton Hospital, Leeds
  - Guy's and St Thomas's NHS Foundation Trust, London
  - Chelsea & Westminster NHS Foundation Trust, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - University of Manchester, Salford
  - Warwick Hospital, Warwick

REFERENCES:
- [Background] Pedro Herranza, Lidia Trasobaresb, Almudena Mateuc, Esperanza Martínezd, Ricardo Ruiz-Villaverdee, Ofelia Baniandrésf, Javier Mataixg, Natalia Jiménez-Gómezh, Marta Serrai, Diana Patricia Ruiz Genaoj, Noelia Riverak, Jesús Tercedor-Sánchezl, Carmen Garciam, Myriam Cordeyn, Enrique Herrera-Acostao. Characterization and outcomes of patients treated with apremilast in the Spanish routine clinical practice: Results from the APPRECIATE study. Actas Dermosifiliogr.
- [Background] Cetkovska P, Dediol I, Sola M, Kojanova M, Trcko K, Carija A, Ceovic R, Ledic-Drvar D, Kastelan M, Hrabar A, Missoup MC, Mamun K. Apremilast Use in Severe Psoriasis: Real-World Data from Central and Eastern Europe. Adv Ther. 2023 Apr;40(4):1787-1802. doi: 10.1007/s12325-023-02468-3. Epub 2023 Mar 2. PMID 36862361
- [Derived] da Silva Burger N, Tran KV, Typou M, Sommer R, Neasham D, Cordey M, Augustin M. Benefits and Satisfaction with Apremilast Treatment in Patients with Psoriasis Affecting the Genital Area: Secondary Analysis of the APPRECIATE Study. Dermatol Ther (Heidelb). 2025 Mar;15(3):681-695. doi: 10.1007/s13555-025-01360-y. Epub 2025 Feb 19. PMID 39969771
- [Derived] Jonak C, Gottfried I, Perl-Convalexius S, Gruber B, Schutz-Bergmayr M, Vujic I, Weger W, Schicher N, Semlin L, Hemetsberger M, Cordey M, Sator P. Characteristics and outcomes of patients with psoriasis treated with apremilast in the real-world in Austria - results the APPRECIATE study. Ther Adv Chronic Dis. 2023 Feb 7;14:20406223231152785. doi: 10.1177/20406223231152785. eCollection 2023. PMID 36777399
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Expanded Access for CC-10004 — https://clinicaltrials.gov/ct2/show/NCT02740218?term=CC-10004-PSOR-013&rank=1